CLINICAL TRIAL: NCT01242800
Title: A Randomized Phase III Trial of the Value of Early Local Therapy for the Intact Primary Tumor in Patients With Metastatic Breast Cancer
Brief Title: Early Surgery or Standard Palliative Therapy in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2108; ECOG-E2108 (Other: ECOG-ACRIN Cancer Research Group); U10CA180794 (NIH)
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Results first posted 2023-02-02 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Stage IV Breast Cancer
Keywords: stage IV breast cancer; local therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): Patients receive standard palliative therapy, if needed, to address symptoms such as tumor ulceration, pain, bulky adenopathy causing arm symptoms, and other similar situations. Therapy may consist of radiotherapy alone, surgery alone, or a combination of both.
  Interventions: Procedure: palliative surgery; Radiation: palliative radiation therapy
- Arm II (Experimental): Patients undergo surgery comprising breast-conserving therapy (BCT) or total mastectomy according to patient and treating physician preference. Surgery is to occur no later than 10 weeks after completion of 32 weeks of systemic therapy. Free surgical margins must be achieved with re-excision or mastectomy for patients undergoing BCT. After completion of BCT, patients undergo radiotherapy once a day, 5 days per week. Patients who had mastectomy undergo radiotherapy at the discretion of treating physician.
  Interventions: Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Procedure: palliative surgery — Undergo standard palliative surgery
  Arms: Arm I
Procedure: therapeutic conventional surgery — Undergo early surgery
  Arms: Arm II
Radiation: palliative radiation therapy — Undergo standard palliative radiotherapy
  Arms: Arm I
Radiation: radiation therapy — Undergo radiotherapy
  Arms: Arm II

SUMMARY:
RATIONALE: The primary tumor might be a source of re-seeding of distant sites and therefore elimination of this source of metastasizing cells by early local therapy may be of benefit.

PURPOSE: This randomized phase III trial is studying early surgery to see how well it works compared to standard palliative therapy in treating patients with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate whether early local therapy of intact primary disease in patients with Stage IV breast cancer whose disease does not progress during initial optimal systemic therapy, will result in prolonged survival, compared to patients who receive local therapy for palliation only.

Secondary

* To compare the time to uncontrolled chest wall disease between patients who receive early local therapy versus patients who receive palliative local therapy.
* To determine whether there is a difference in health-related quality-of-life (HRQOL) between patients who receive early local therapy versus patients who receive palliative local therapy.
* To determine whether the absolute value of circulating tumor cells (CTC) burden at 6 months following randomization (time +6) will be lower in the palliative therapy arm than in early local therapy arm, and whether this value is inversely related to survival (lower CTC, longer survival).

Exploratory

* To collect tumor and blood specimens for future exploration of the biological interactions between the primary tumor and metastatic lesions and the effect of primary tumor resection.

OUTLINE: This is a multicenter study. Patients are stratified according to hormone receptor and treatment plan (ER+ or PR+, HER2-, endocrine therapy alone vs ER+ or PR+, and HER2-, chemotherapy and/or endocrine therapy vs ER- or PR-, and HER2- vs HER2+), and number of involved organ systems with distant disease (regional nodes in the axillary, supraclavicular, and internal mammary locations are not considered distant sites) (1 vs > 1). Patients are randomized to 1 of 2 treatment arms in 1:1 ratio.

* Arm I: Patients receive standard palliative therapy, if needed, to address symptoms such as tumor ulceration, pain, bulky adenopathy causing arm symptoms, and other similar situations. Therapy may consist of radiotherapy alone, surgery alone, or a combination of both.
* Arm II: Patients undergo surgery comprising breast-conserving therapy (BCT) or total mastectomy according to patient and treating physician preference. Surgery is to occur no later than 10 weeks after completion of 32 weeks of systemic therapy. Free surgical margins must be achieved with re-excision or mastectomy for patients undergoing BCT. After completion of BCT, patients undergo radiotherapy once a day, 5 days per week. Patients who had mastectomy undergo radiotherapy at the discretion of treating physician.

Patients may undergo blood and tumor tissue sample collection for circulating tumor cells (CTC) burden and future studies.

Patients complete the Functional Assessment of Cancer Therapy - Breast Trial Outcome Index (FACT- TOI) and FACT - General (22) and the Breast Cancer Subscale (FACT-B) quality-of-life questionnaires at baseline and periodically during study.

After completion of study therapy, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intact primary (not recurrent) invasive carcinoma of the breast

  * Stage IV disease
  * Confirmation of the primary tumor should be by needle biopsy (preferred)
  * Incisional surgical biopsy allowed as long as there is residual palpable or tumor image in the breast
* Patients must be judged to be candidates for complete resection with free margins followed by radiation therapy (if radiation therapy is indicated)
* For women not undergoing axillary dissection, sentinel node biopsy should document an axillary nodal burden of 1-2 involved lymph nodes (i.e., ACOSOG Z-11 criteria may be applied)
* Prior non-invasive (Ductal Carcinoma In Situ) cancer allowed provided there has been no recurrence
* Prior ipsilateral invasive cancer allowed if more than 5 years previous
* Patients should have at least one organ system involved with distant metastatic disease

  * If patient has only one metastatic lesion/focus, this must be proven by biopsy and the pathology report confirming the diagnosis of primary breast cancer, as well as the metastatic site, must be available
* Must have available radiologic reports documenting disease status within the past 6 weeks prior to initiating systemic therapy
* CNS metastases allowed provided projected survival > 6 months
* Patients must have completed at least 16 weeks of optimal systemic therapy (appropriate to the tumor biological profile and the patient's age and menopausal status)

  * If systemic therapy is discontinued for toxicity, but there is no distant progression and at least 12 weeks of therapy have been delivered, then the patient remains eligible
  * Radiation therapy (if indicated) must begin within 12 weeks of final therapeutic surgical procedure (including re-excision for free margins and completion of axillary dissection)
* Patients may register at any time from the time of diagnosis of stage IV breast cancer (if eligibility criteria met) to the time when a maximum of 30 weeks of induction systemic therapy has been completed

  * Patients must be randomized within 16-32 weeks after the start of systemic therapy
* Patients must not have experienced disease progression since the start of systemic therapy, as evidenced by radiographic documentation of disease status before treatment and within 4 weeks +/- 2 weeks prior to randomization, including:

  * No new sites of disease
  * No enlargement of existing sites by 20% or more in longest diameter
  * No symptomatic deterioration
* Patients who require radiotherapy to bone metastases during induction systemic therapy are eligible
* Local disease at the primary site must be asymptomatic
* Hormone receptor status known
* Menopausal status not specified
* Patients must have adequate organ function to undergo local therapy 4 weeks +/- 2 weeks prior to randomization per investigator discretion and institutional guidelines
* More than 5 years since other primary cancers that were curatively treated
* Negative pregnancy test
* Fertile patients must use an accepted and effective contraception method

Exclusion criteria:

* Synchronous contralateral breast cancer
* Pregnant or nursing

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2011-05-16 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema A. Khan, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (377):
- United States (369):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - North Bay Cancer Center, Fairfield, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Community Hospital of the Monterey Peninsula Comprehensive Cancer Center, Monterey, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Stanford Cancer Center, Stanford, California
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Leeward Radiation Oncology, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute, Nampa, Idaho
  - Mountain States Tumor Institute at St. Luke's, Twin Falls, Idaho
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center at Catholic Medical Center, Manchester, New Hampshire
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Radiation Oncology Center at Kennedy Health System - Sewell, Sewell, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Winthrop University Hospital, Mineola, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Dyson Center for Cancer Care at Vassar Brothers Medical Center, Poughkeepsie, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Charles A. & Betty Bott Cancer Center at Holy Redeemer Hospital, Meadowbrook, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Baylor Medical Center at Irving, Irving, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - St. Mary Regional Cancer Center at St. Mary Medical Center, Walla Walla, Washington
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Fox Valley Surgical Associates at Appleton Medical Center, Appleton, Wisconsin
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
- Canada (5):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia
- Pretoria Academic Hospital, Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Khan SA, Zhao F, Goldstein LJ, Cella D, Basik M, Golshan M, Julian TB, Pockaj BA, Lee CA, Razaq W, Sparano JA, Babiera GV, Dy IA, Jain S, Silverman P, Fisher CS, Tevaarwerk AJ, Wagner LI, Sledge GW. Early Local Therapy for the Primary Site in De Novo Stage IV Breast Cancer: Results of a Randomized Clinical Trial (EA2108). J Clin Oncol. 2022 Mar 20;40(9):978-987. doi: 10.1200/JCO.21.02006. Epub 2022 Jan 7. Erratum In: J Clin Oncol. 2022 Apr 20;40(12):1392. doi: 10.1200/JCO.22.00666. PMID 34995128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on February 8, 2011, accrued its first patient on May 16, 2011, and accrual was terminated on July 23, 2015 with a final accrual of 390 patients on Step 1. Of the 390 patients enrolled, 256 of them were randomized to Step 2 to arm I and arm II.
Groups:
- Arm I (Continued Systemic Therapy): Patients receive standard palliative therapy, if needed, to address symptoms such as tumor ulceration, pain, bulky adenopathy causing arm symptoms, and other similar situations. Therapy may consist of radiotherapy alone, surgery alone, or a combination of both.
  palliative surgery: Undergo standard palliative surgery
  palliative radiation therapy: Undergo standard palliative radiotherapy
- Arm II (Early Local Therapy): Patients undergo surgery comprising breast-conserving therapy (BCT) or total mastectomy according to patient and treating physician preference. Surgery is to occur no later than 10 weeks after completion of 32 weeks of systemic therapy. Free surgical margins must be achieved with re-excision or mastectomy for patients undergoing BCT. After completion of BCT, patients undergo radiotherapy once a day, 5 days per week. Patients who had mastectomy undergo radiotherapy at the discretion of treating physician.
  therapeutic conventional surgery: Undergo early surgery
  radiation therapy: Undergo radiotherapy
Period: Overall Study
Arm/Group | Arm I (Continued Systemic Therapy) | Arm II (Early Local Therapy)
Started | 131 | 125
Completed | 131 (Patient continued their systemic therapy after randomization per their treating physician's discretion.) | 106 (Protocol therapy was early surgery and/or radiation therapy in this trial.)
Not Completed | 0 | 19
Not completed — Patient refusal | 0 | 10
Not completed — Physician Decision | 0 | 1
Not completed — Disease progression | 0 | 3
Not completed — Lack of insurance coverage for surgery | 0 | 1
Not completed — Reasons not reported | 0 | 4

BASELINE CHARACTERISTICS:
Population: All randomized patients at step 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Continued Systemic Therapy) | Arm II (Early Local Therapy) | Total
Number analyzed (Participants) | 131 | 125 | 256
Age, Continuous [Median (Full Range); unit: years] | 56 [25 to 86] | 55 [30 to 81] | 56 [25 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 125 | 256
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 19 | 19 | 38
  White | 102 | 98 | 200
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: 3-year Overall Survival Rate
Description: Overall survival (OS) was defined as time from randomization to death from any cause. All patients will be followed for survival through 5 years. Cases with incomplete follow-up or without record of vital status will be censored at the date of last contact. 3-year OS rate was estimated using Kaplan-Meier method.
Time Frame: Assessed at baseline, then every 3 months within 2 years and every 6 months between 2-5 years, up to 5 years
Population: All randomized patients at step 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Continued Systemic Therapy) | Arm II (Early Local Therapy)
Number analyzed (Participants) | 131 | 125
percentage of participants | 67.9 [58.8 to 75.5] | 68.4 [59.0 to 76.1]
Statistical Analysis 1: Comparison: Arm I (Continued Systemic Therapy) vs Arm II (Early Local Therapy); Test type: Superiority; p = 0.32, Log Rank; Stratified log rank test was used for arm comparison

2. Secondary Outcome: 3-year Cumulative Incidence of Locoregional Recurrence/Progression
Description: For patients in arm II (early local therapy), time to locoregional recurrence was defined as time from randomization to date of locoregional recurrence; for patients in arm A (continued systemic therapy), time to locoregional progression was defined as time from randomization to date of locoregional progression. In this study, locoregional recurrence was defined as the new development or clinically significant increase in size of any supraclavicular, infraclavicular, internal mammary or axillary adenopathy or chest wall disease or invasive in-breast recurrence for patients on arm B; for patients on arm A, locoregional progression was defined as the development of symptoms leading to a decision for local therapy. Locoregional recurrence/progression and distant progression were followed separately in the study, and the occurrence of one did not preclude the other getting reported. 3-year cumulative incidence of locoregional recurrence/progression was estimated.
Time Frame: Assessed at baseline, then every 3 months within 2 years and every 6 months between 2-5 years, up to 5 years
Population: All randomized patients at step 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Continued Systemic Therapy) | Arm II (Early Local Therapy)
Number analyzed (Participants) | 131 | 125
percentage of participants | 16.3 [10.7 to 24.4] | 39.8 [31.8 to 49.1]

3. Secondary Outcome: Health-related Quality of Life (HRQL)
Description: The Functional Assessment of Cancer Therapy-Breast Trial Outcome Index (FACT-B TOI) was used as the primary HRQL endpoint, measured by the prorated aggregate score of the 24 items from the FACT-B (7 functional well-being, 7 physical well-being, 10 breast cancer specific items). The theoretical range of the prorated aggregate score was 0-96, higher scores indicate better quality of life.
Time Frame: Assessed at 18 months after randomization
Population: All randomized patients at step 2 who reported quality of life data at 18 months after randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Continued Systemic Therapy) | Arm II (Early Local Therapy)
Number analyzed (Participants) | 65 | 66
score on a scale | 74.2 (11.5) | 68.0 (13.7)

ADVERSE EVENTS:
Time Frame: The trial involved standard of care systemic therapies and there could be many options of systemic therapies, adverse events data were not collected in the trial. For all-cause mortality, it was assessed every 3 months within 2 years and every 6 months between 2-5 years, up to 5 years.
Description: The trial involved standard of care systemic therapies and there could be several options of systemic therapies, adverse events data were not collected in the trial.
Arm/Group | Arm I (Continued Systemic Therapy) | Arm II (Early Local Therapy)
All-Cause Mortality (participants affected / at risk) | 63/131 | 58/125
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT01242800/Prot_SAP_000.pdf